CLINICAL TRIAL: NCT02497456
Title: The Effectiveness of a Counselling Intervention on the Uptake of HIV Care Services Among HIV Infected Patients in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Linkage to pre-ART care
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: HIV
Keywords: HIV; Counselling; Care; antiretroviral therapy; linkage; Uganda; Africa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow-up counselling (Experimental): Participants in the experimental arm will receive home-based HIV counselling and testing and referral for HIV care if found to have HIV infection. Additionally, participants will receive home-based follow-up counselling at 1 and 2 months after HIV diagnosis.
  Interventions: Behavioral: Follow-up counselling
- Standard of care (No Intervention): Participants in this arm will receive only home-based HIV counselling and testing and referral for HIV care if found to have HIV infection.

INTERVENTIONS:
Behavioral: Follow-up counselling
  Arms: Follow-up counselling

SUMMARY:
The purpose of this study is to evaluate the impact of follow-up counselling after HIV diagnosis through home-based HIV counselling and testing (HBHCT), on linkage to pre-antiretroviral therapy (pre-ART) care in Uganda.

DETAILED DESCRIPTION:
Data on linkage to pre-antiretroviral therapy (pre-ART) care after HIV diagnosis through home-based HIV counselling and testing (HBHCT) in sub-Saharan Africa (SSA) are scarce. The few existing data suggest that only 13% to 54% of HIV-infected persons identified through HBHCT enter pre-ART care. No studies have rigorously evaluated interventions aimed at improving linkage to pre-ART care following HBHCT in SSA. This study will evaluate the effect of follow-up counselling after HIV diagnosis through HBHCT on linkage to pre-ART care in Masaka, south-western Uganda.

The study is a cluster randomised trial of the effectiveness of referral to pre-ART care and follow-up counselling (intervention) compared to referral to pre-ART care only (control), for individuals diagnosed with HIV through HBHCT. The intervention will be administered at months 1 and 2, and linkage to care assessed at month 6 post-HBHCT. Data will be collected on socio-demographic characteristics, sexual risk profile, HIV testing history, HIV status disclosure, linkage to care, CD4 count testing and results, cotrimoxazole prophylaxis, and ART initiation. At least 224 HIV-infected participants will be enrolled from 28 clusters (14/study arm). Approximately 84 HIV-uninfected individuals will also be recruited into the study to reduce the possibility of revealing the sero-status of the HIV-infected participants.

ELIGIBILITY:
HIV-infected participants

Inclusion Criteria:

1. HIV-infected adult (≥18 years)
2. Willing to provide informed consent
3. Willing to receive follow-up counselling at home

Exclusion Criteria:

1. Previous or current receipt of HIV care from an ART provider
2. On-going participation in other health-related research
3. Intending to change residence in the next 6 months
4. Conditions that may make it difficult to provide informed consent e.g. reported (by the individual, relatives or other community members) on-going psychiatric illness

HIV-uninfected participants

Inclusion criteria:

1. HIV negative adult (≥18 years)
2. Willing to provide informed consent
3. Willing to receive follow-up counselling at home

Exclusion criteria:

1. Intending to change residence in the next 6 months
2. Conditions that may make it difficult to provide informed consent e.g. reported (by the individual, relatives or other community members) on-going psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The proportion of HIV-infected participants that register with an anti-retroviral therapy (ART) care provider within 3 and 6 months of HIV diagnosis and referral. | 6 months
The time between HIV diagnosis and linkage to pre-ART care. | 6 months

SECONDARY OUTCOMES:
Time between blood draw for CD4 cell count testing and attending clinic to receive the results among participants that link to pre-ART care | 6 months
The time between learning that a participant is eligible for ART and ART initiation | 6 months
The proportion of participants who report adherence to daily cotrimoxazole prophylaxis at 3 and 6 months after HIV diagnosis through HBHCT among those that link to pre-ART care. | 6 months

OTHER OUTCOMES:
The proportion of individuals who undergo repeat HIV testing within 6 months of testing HIV negative through HBHCT. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Ruzagira, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit
Locations (1):
- MRC/UVRI Uganda Research Unit on Aids, Masaka, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruzagira E, Grosskurth H, Kamali A, Baisley K. Brief counselling after home-based HIV counselling and testing strongly increases linkage to care: a cluster-randomized trial in Uganda. J Int AIDS Soc. 2017 Oct;20(2):e25014. doi: 10.1002/jia2.25014. PMID 29052344